CLINICAL TRIAL: NCT01126697
Title: PITT0908: Clinical Trial of Coenzyme Q10 and Lisinopril in Muscular Dystrophies
Brief Title: Clinical Trial of Coenzyme Q10 and Lisinopril in Muscular Dystrophies
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PITT0908
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Limb Girdle Muscular Dystrophy
Keywords: Cardiac; Muscular Dystrophy; Randomized
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies, Limb-Girdle; Muscular Dystrophies | interventions — coenzyme Q10; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Enhanced standard of care (No Intervention)
- Lisinopril (Active Comparator)
  Interventions: Drug: Coenzyme Q10 and Lisinopril
- Coenzyme Q10 (Active Comparator)
  Interventions: Drug: Coenzyme Q10 and Lisinopril
- Coenzyme Q10 and Lisinopril (Active Comparator)
  Interventions: Drug: Coenzyme Q10 and Lisinopril

INTERVENTIONS:
Drug: Coenzyme Q10 and Lisinopril — Arm 1. Coenzyme Q10: taken once a day each morning by mouth OR Arm 2. Lisinopril: taken once a day each morning by mouth OR Arm 3. Coenzyme Q10 and lisinopril: each taken once a day in the morning by mouth OR Arm 4. Enhanced Standard Care (more doctor visits, muscle and breathing testing, and x-rays for monitoring, but no study medication).
  Arms: Coenzyme Q10; Coenzyme Q10 and Lisinopril; Lisinopril

SUMMARY:
The study will include 120 participants aged 8 and up with Duchenne, Becker, or autosomal recessive limb-girdle (specifically: LGMD 2C-2F and 2I) muscular dystrophies that have no clinical cardiac symptoms. Participants will be randomized to one of four arms: Arm 1 CoQ10 alone, Arm 2 Lisinopril alone, Arm 3 CoQ10 and Lisinopril or Arm 4 No study medication. Randomization will be stratified by ambulatory status and corticosteroid use. The primary outcome for the study is the myocardial performance index (MPI), measured by standard Doppler echocardiography. The study will last 24 months with visits at Months 0.5,1.5, 6, 12, 18 and 24.

Following completion of the Clinical Trial of Coenzyme Q10 and Lisinopril, participants will be offered participation in a companion protocol: PITT1215 A Natural History Companion Study to PITT0908: Clinical Trial of Coenzyme Q10 and Lisinopril in Muscular Dystrophies. The objective of this study is to evaluate the longitudinal natural history of DMD, BMD, and LGMD2I and to evaluate the effects of Coenzyme Q10 and/or Lisinopril on prevention of cardiac dysfunction in these disorders.This will be an 18-month longitudinal natural history study designed to accompany the Clinical Trial of Coenzyme Q10 and Lisinopril in Muscular Dystrophies.

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age or older
* Confirmed genetic diagnosis of Duchenne, Becker, or Limb Girdle muscular dystrophy
* Beta-blocker naïve
* Screening Doppler echocardiographic MPI measurement greater than or equal to 0.40 for the highest MPI value (spectral and tissue) or circumferential strain measured by STE that is less negative than or equal to - 23
* Normal left ventricular fractional shortening (≥28%) and no clinical cardiac symptoms
* Has not participated in other therapeutic research protocol within the last 6 months prior to screening
* Ability to swallow tablets

Exclusion Criteria:

* Spine curvature greater than 30% (based on the x-ray performed at screening)
* History of significant concomitant illness or significant impairment of renal or hepatic function
* History of hypersensitivity to ACE inhibitors
* History of idiopathic or hereditary angioedema or a history of angioedema with prior ACE inhibitor use
* Use of carnitine, creatine, glutamine, or any herbal medicines (this would not include herbal teas unless they are consumed daily with intended medicinal effect) in the 3-months prior to enrollment
* CoQ10 and/or ACE inhibitor use for a duration greater than 6 months
* CoQ10 and/or ACE inhibitor use in the 3-months prior to enrollment
* CoQ10 serum level of 2.5 ug/ml or higher
* Investigator assessment of inability to comply with protocol

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
myocardial performance index (MPI) | every 6 months
  The MPI is a sensitive, quantifiable, noninvasive measure of global ventricular function that is independent of cardiac geometry and heart rate. MPI is collected through standard echocardiogram assessment. MPI is a ratio of the total time spent in isovolumic activity (isovolumic contraction time and isovolumic relaxation time) to the time spent in ventricular ejection.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital, Chicago, Illinois
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
- Alberta Children's Hospital, Calgary, Alberta, Canada
- National Center of Neurology and Psychiatry, Tokyo, Japan

REFERENCES:
- See also: CINRG Network Website — http://www.cinrgresearch.org